CLINICAL TRIAL: NCT07155590
Title: Subphenotype- and Complication-guided Adjunctive Fosfomycin Therapy for Staphylococcus Aureus Bacteraemia: Pooled Analysis of Two Randomised Trials
Brief Title: Subphenotype- and Complication-guided Adjunctive Fosfomycin Therapy for Staphylococcus Aureus Bacteraemia
Status: Active, not recruiting | Type: Observational
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); University of Barcelona (Other); Hospital Universitario Virgen Macarena (Other); University of Seville (Other)
Responsible Party: Principal Investigator, Francesc Escrihuela-Vidal, MD, PhD, Hospital Universitari de Bellvitge
Other Study IDs: FENAUREUS-BACSAFO
Record Dates: First submitted 2025-08-27; First posted 2025-09-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Staphylococcal Aureus Infection; Staphylococcus Aureus Bacteraemia
Keywords: Staphylococcus aureus bacteraemia; Risk stratification; Clinical phenotypes; Subphenotypes; Monotherapy; Adjunctive therapy; Fosfomycin; Complicated bacteraemia; Randomised clinical trials

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adjunctive fosfomycin therapy: Patients with Staphylococcus aureus bacteraemia from the BACSAFO cohort treated with any regimen including fosfomycin
- Monotherapy: Patients with Staphylococcus aureus bacteraemia from the BACSAFO cohort treated with any regimen not containing fosfomycin

SUMMARY:
Staphylococcus aureus bacteraemia (SAB) is a major global cause of sepsis-related mortality. Randomised trials of adjunctive antibiotics, including fosfomycin, have not shown consistent benefit, possibly due to inclusion of unselected SAB populations. The FEN-AUREUS classification enables early risk stratification based on clinical subphenotypes. The investigators aim to validate this framework in a pooled trial cohort and assess whether combining subphenotypes with IDSA-defined complicated SAB could identify patients most likely to benefit from adjunctive fosfomycin. The investigators will conduct a post-hoc analysis of individual-level data from two multicentre randomised trials-BACSARM and SAFO-evaluating fosfomycin in SAB. Participants will be classified using FEN-AUREUS into source phenotypes (A, B and C) and risk subphenotypes (1 = low-risk, 2 = high-risk). Associations between subphenotype, treatment arm, and outcomes (30/60-day mortality, 8-week treatment success) will be assessed using multivariable models. Monte Carlo simulations will explore power by subgroup. FEN-AUREUS subphenotypes combined with complication status have the potential to identify patients with SAB that could likely benefit form combination therapy with fosfomycin.

ELIGIBILITY:
Inclusion criteria for the present study: all patients included in the BACSAFO cohort, composed of all patients included in the intention-to-treat populations of the BACSARM and SAFO randomised clinical trials (RCT).

Inclusion criteria for the BACSARM and SAFO RCTs:

* > or = 18 years old
* Monomicrobial Staphylococcus aureus bacteraemia
* Evidence of active infection

Common exclusion criteria for the BACSARM and SAFO RCTs:

* Polymicrobial bacteraemia
* Severe clinical status with expected survival < 24 hours
* Severe liver disease with Child-Pugh score class C
* Diagnosis of prosthetic infective endocarditis
* Allergy or known resistance to study drugs
* Pregnancy at the time of inclusion
* Inclusion in another clinical trial

Particular exclusion criteria for the BACSARM RCT:

* Diagnosis of MRSA pneumonia
* Prior history of eosinophilic pneumonia
* Use of additional antibiotic therapy with microbiological activity against MRSA

Particular exclusion criteria for the SAFO RCT:

* Prior history of myasthenia gravis
* Acute SARS-CoV2 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The BACSAFO cohort pools individual participant data from two multicentre, randomised, superiority trials evaluating adjunctive fosfomycin for the treatment of SAB: BACSARM and SAFO. The BACSARM trial included 155 adult patients with methicillin-resistant (MRSA), randomised 1:1 to receive either daptomycin alone or daptomycin plus fosfomycin. The SAFO trial enrolled 214 adult patients with methicillin-susceptible (MSSA) bacteraemia, randomised to cloxacillin alone or cloxacillin plus fosfomycin.
Sampling Method: Probability Sample
Enrollment: 369 (Actual)
Dates: Start 2025-07-21 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 60 days | At 60 days from randomisation
  All-cause mortality at 60 days after randomisation

SECONDARY OUTCOMES:
All-cause mortality at 30 days | At 30 days after randomisation
  All-cause mortality at 30 days after randomisation
Treatment success at 8 weeks | At 8 weeks after randomisation
  Survival without clinical relapse and with resolution of symptoms at 8 weeks after randomisation

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Universitario Virgen de Macarena, Seville

IPD SHARING:
Plan to Share IPD: Yes
Raw anonymised data relating to primary and secondary outcomes and safety may be shared upon request with researchers who provide a methodologically reasonable proposal. Requests for data should be sent to the corresponding author (JC). Interested researchers must obtain the approval of the Bellvitge University Hospital Ethics Committee.
Supporting Information: Study Protocol, SAP, CSR